CLINICAL TRIAL: NCT03069976
Title: " Overlap Syndrome and PSC: Evaluating Role of Gut Microflora and Its Modification With Antibiotics in Children"
Brief Title: "Overlap Syndrome and PSC: Evaluating Role of Gut Microflora and Its Identification With Antibiotics in Children"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OS.ABBA.CH.1618
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Primary Sclerosing Cholangitis; Autoimmune Hepatitis; Overlap Syndrome
MeSH Terms: conditions — Cholangitis, Sclerosing; Hepatitis, Autoimmune | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All included patients, diagnosed with Overlap Syndrome or Primary Sclerosing Cholangitis, will receive treatment (Metronidazole x 14 days) hence single arm study.
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Metronidazole — Flagyl x 14 days.
  Other Names: Flagyl

SUMMARY:
Based upon the possible implication of microbiota and abnormal microbial metabolites such as altered bile acids, in the pathogenesis of PSC, emerging data suggests that oral antibiotics, such as vancomycin and metronidazole, may have therapeutic effects in this overlap syndrome or PSC.

The goal of our study is to evaluate role of antibiotics and microflora in children with AIH/PSC overlap syndrome or with PSC alone. The investigators hope to learn what effects oral antibiotics has on the bacteria present in stool, and hope to learn to characterize human intestinal microbial communities, in children suffering from overlap syndrome or PSC.

The hypothesis of the investigators is that overlap syndrome and PSC develop due to altered microflora and the resulting abnormal bile acids pool. The outcome of overlap syndrome or PSC could be affected by presence or absence of RCUH. Antibiotics to correct the microflora may result in disease/cholangiopathy remission.

DETAILED DESCRIPTION:
The used antibiotic is Metronidazole (Flagyl), during 14 days, as induction therapy or rescue therapy.

Study participants will provide blood and stool samples in order to evaluate bile acids profile and microbiome, before and after the course of metronidazole, and then comparison will be made pre- and post-antibiotics.

The investigators will determine the benefit of oral metronidazole therapy through improvement of clinical symptoms and improvement of liver function tests.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with overlap syndrome, overlap syndrome + ulcerative colitis (UC), Primary sclerosing cholangitis (PSC) or PSC + UC
* Children for whom consent is available
* Children under regular follow-up
* Children with at least one liver biopsy (for overlap syndrome patients)
* Children with at least one liver biopsy and one MRCP (for PSC patients)

Exclusion Criteria:

* Death
* Patients older than 18 years old at the time of diagnosis of liver disease

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01; Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Liver function test | 14 days
  AST, ALT, GGT to be measured

SECONDARY OUTCOMES:
Microbiome | 14 days
  Intestinal microflora to be characterized
Bile acid profile | 14 days
  Bile acids profile to be characterized

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Sokal, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc - Université Catholique de Louvain, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No